CLINICAL TRIAL: NCT00628914
Title: Brain Mechanisms and Targeting Insomnia in Major Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Ian A. Cook, M.D., University of California Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESRC973; 07-11-013
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-07

CONDITIONS: Major Depressive Disorder; Insomnia
Keywords: Major Depressive Disorder; Insomnia; Escitalopram; Lexapro; Eszopiclone; Lunesta; Cordance
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — Escitalopram; Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Open label escitalopram plus eszopiclone for 8 weeks
  Interventions: Drug: escitalopram and eszopiclone
- 2 (Other): Escitalopram and eszopiclone for initial 4 weeks, then switch to escitalopram and placebo for final 4 weeks.
  Interventions: Drug: Escitalopram, eszopiclone, and placebo
- 3 (Placebo Comparator): Escitalopram plus placebo for 8 weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: escitalopram and eszopiclone — escitalopram 10mg tabs QD and eszopiclone 3 mg tabs QD for 8 weeks
  Other Names: Lexapro; Lunesta
  Arms: 1
Drug: Escitalopram, eszopiclone, and placebo — Escitalopram 10mg tabs QD for 8 weeks; Eszopiclone 3mg tabs QD for initial 4 weeks then placebo tabs QD for final 4 weeks
  Other Names: Lexapro; Lunesta
  Arms: 2
Drug: Escitalopram — Escitalopram 10mg tabs QD and placebo tabs QD for 8 weeks
  Other Names: Lexapro
  Arms: 3

SUMMARY:
Preliminary studies suggest that the response to antidepressant medication can be accelerated by targeting insomnia with adjunctive use of eszopiclone. It is not yet known what mechanism(s) support this acceleration in response, though preliminary findings support the hypothesis that early restoration of sleep may facilitate BDNF-based effects of antidepressant medications. The optimal duration of co-treatment is also unknown. This study will test specific hypotheses about brain mechanisms and evaluate the effects of continued eszopiclone beyond the time window when response acceleration should be observed.

DETAILED DESCRIPTION:
A critical challenge in the management of major depressive disorder (MDD) is the delay between initiating treatment with an antidepressant medication and clinical improvement. Preliminary studies (Fava et al., 2006; Krystal et al., 2007) suggest that targeting insomnia with eszopiclone (ESZ) in patients receiving fluoxetine may lead to more rapid resolution of symptoms. Studies have not yet been able to differentiate between competing explanations of this phenomenon: whether co-treatment with ESZ actually accelerates changes in the brain associated with antidepressant treatment response, or if its effects on the insomnia component are confined to the symptomatic level ("masking"). As a non-benzodiazepine GABA-receptor agonist with FDA approval for long-term use in the treatment of sleep disturbances, ESZ is an appropriate agent for targeting insomnia in MDD without major concerns around the development of tolerance. Further research in co-treatment would be advanced by understanding the mechanism(s) underlying accelerated improvement.

Our prior work (Cook et al., 2001, 2002, 2005; Leuchter et al. 2002) has studied a new physiologic biomarker of response to SSRI and mixed-action antidepressants. The EEG-based cordance biomarker can detect the physiologic effects of successful antidepressant treatment at 48 hours, 1 week, and 2 weeks of treatment; in contrast, symptom differences between responders and non-responders did not separate until 4 weeks of treatment in our placebo-controlled trials. Additionally, the magnitude of early physiologic change was associated with the completeness of clinical response. Our biomarker has been independently studied and our findings replicated (Bareš et al., 2007). The cordance biomarker can be considered as a leading indicator or predictor of treatment outcome. As a non-invasive probe of brain physiology, it may detect early neurophysiologic changes associated with accelerated clinical response from eszopiclone.

Other research has reported that brain derived neurotrophic factor (BDNF) is reduced in many patients with MDD (Karege et al., 2002, 2005, Shimizu et al., 2003) and may rise during the course of treatment with antidepressant medication (e.g., Gonul et al., 2005; Yoshimura et al., 2007; Huang et al., 2007). BDNF-related neuroplasticity has been suggested as a mechanism by which medications can lead to mood improvement (Duman 2002; Manji et al., 2003). Sleep patterns have also been shown to have an impact on neuroplasticity (Taishi et al., 2001; cf. Benington & Frank, 2003). A simple acute phase-shift in sleep can impact BDNF levels (Sei 2003), suggesting that a link between sleep and symptomatic recovery from depression might operate via a BDNF mechanism and reflect changes in brain physiology.

While Krystal and colleagues (2007) previously reported that the beneficial clinical effects of 8 weeks of co-treatment did not diminish significantly in the two weeks following ESZ discontinuation, controlled studies have not examined outcomes in clinically-likely scenarios employing shorter co-treatment periods (e.g., 4 weeks, during which much of the acceleration occurs).

Based on these previous studies, this study will assess patients with MDD during treatment with an SSRI antidepressant, escitalopram (ESC), administered along with either ESZ or placebo (PBO), using (a) clinical symptom ratings, (b) serum levels of BDNF, (c) cognitive function, and (d) brain physiology with EEG.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with non-psychotic, unipolar Major Depressive Disorder (MDD).
* A score of >14 on the HAM-D17.
* Presence of insomnia, manifest by a total score of ≥ 4 combining all three sleep disturbance items on the HAM-D17 scale.
* Age range: 18-64.
* Patients with suicidal ideation are eligible only if the thoughts of death or of life not being worth living are not accompanied by a plan or intention for self-harm.

Exclusion Criteria:

* Patient is mentally or legally incapacitated, unable to give informed consent.
* Patients who have a lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, MDD with psychotic features, or dementia (any etiology).
* Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
* Patients with a current diagnosis of anorexia nervosa, bulimia nervosa, or obsessive compulsive disorder.
* Patients who have met diagnostic criteria for any current substance abuse disorder at any time in the 6 months prior to enrollment.
* Insomnia symptoms that have not responded to a previous trial of a sedativehypnotic prescription medication.
* Any history of seizures, brain surgery, skull fracture, significant head trauma, or previous abnormal EEG.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-11 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Change in cordance value | Visits 2-9
Change in cordance value | Visit 11
Change in cordance value | Visit 13

SECONDARY OUTCOMES:
Depression symptom severity | each visit
Serum BDNF | visits 2-9
Cognitive testing | visits 2-7
Serum BDNF | Visit 11
Serum BDNF | Visit 13
Cognitive testing | Visit 9
Cognitive testing | Visit 13

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, MD, Principal Investigator — Semel Institute for Neuroscience and Human Behavior at UCLA
Locations (1):
- Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California, United States

REFERENCES:
- See also: UCLA Depression Research Program — http://www.DepressionLA.com/
- See also: UCLA Laboratory of Brain, Behavior, and Pharmacology — http://www.lbbp.org/